CLINICAL TRIAL: NCT04859296
Title: Analgesic and Appetite-stimulating Effects of Cannabigerol Administered Alone and in Combination With Delta-9-tetrahydrocannabinol
Brief Title: AnalgeSiC and appEtite-stimulating Effects of caNnabigerol and THC (ASCENT)
Acronym: ASCENT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-000208
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Pain; Appetite Loss; Abuse, Drug
Keywords: Analgesia; Pain; Appetite; THC; Cannabigerol; CBG
MeSH Terms: conditions — Pain; Anorexia; Substance-Related Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Placebo (Placebo Comparator): 0 mg CBG, 0 mg THC
  Interventions: Drug: Placebo
- Low strength CBG (Active Comparator): 5 mg CBG, 0 mg THC
  Interventions: Drug: Low CBG
- High strength CBG (Active Comparator): 15 mg CBG, 0 mg THC
  Interventions: Drug: High CBG
- Low strength THC (Active Comparator): 0 mg CBG, 5 mg THC
  Interventions: Drug: Low THC
- High strength THC (Active Comparator): 0 mg CBG, 30 mg THC
  Interventions: Drug: High THC
- Low strength CBG + Low strength THC (Active Comparator): 5 mg CBG + 5 mg THC
  Interventions: Drug: Low CBG; Drug: Low THC
- Low strength CBG + High strength THC (Active Comparator): 5 mg CBG + 15 mg THC
  Interventions: Drug: Low CBG; Drug: High THC
- High strength CBG + Low strength THC (Active Comparator): 15 mg CBG + 5 mg THC
  Interventions: Drug: High CBG; Drug: Low THC
- High strength CBG + High strength THC (Active Comparator): 15 mg CBG + 15 mg THC
  Interventions: Drug: High CBG; Drug: High THC

INTERVENTIONS:
Drug: Placebo — Vaporized placebo
  Arms: Placebo
Drug: Low CBG — Vaporized CBG (5 mg)
  Arms: Low strength CBG; Low strength CBG + High strength THC; Low strength CBG + Low strength THC
Drug: High CBG — Vaporized CBG (15 mg)
  Arms: High strength CBG; High strength CBG + High strength THC; High strength CBG + Low strength THC
Drug: Low THC — Vaporized THC (5 mg)
  Arms: High strength CBG + Low strength THC; Low strength CBG + Low strength THC; Low strength THC
Drug: High THC — Vaporized THC (15 mg)
  Arms: High strength CBG + High strength THC; High strength THC; Low strength CBG + High strength THC

SUMMARY:
This study will assess the analgesic, appetite-stimulating, and subjective effects of cannabigerol (CBG) alone and in combination with THC.

DETAILED DESCRIPTION:
The overall aim of this double-blind, placebo-controlled, within-subject study in healthy, occasional cannabis smokers is to ascertain the dose-dependent analgesic and appetite-stimulating effects of ecologically relevant doses of cannabigerol (CBG) alone and in combination with a sub-analgesic / sub-appetite stimulating, minimally psychoactive dose of THC and an analgesic, appetite-stimulating, but intoxicating dose of THC.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating females aged 21-55 years
* • Report occasional use of cannabis (cannabis use between ≥ biweekly and ≤ 3 days per week) over the month prior to screening
* Not currently seeking treatment for their cannabis use
* Have a Body Mass Index from 18.5 - 34kg/m2.
* Able to perform all study procedures
* Must be using a contraceptive (hormonal or barrier methods)
* Females must not be lactating

Exclusion Criteria:

* Meeting DSM-V criteria for moderate-severe Cannabis Use disorder (CUD) or any substance use disorder other than nicotine, caffeine, or mild CUD
* Any other Axis I disorder
* • Current use of any medications within 14 days or 5 half-lives of administration (whichever is longer) except for hormonal contraceptives in females. If a medication is taken once a participant is enrolled, sessions will be suspended for 14 days or 5 half-lives after administration (whichever is longer)
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process are not within the normal range and / or reveal any significant illness (e.g., hypertension) as judged by the study physician and to put the participant at greater risk of experiencing adverse events due to completion of study procedures.
* Current pain
* Pregnancy is exclusionary due to the possible effects of the study medication on fetal development.
* History of an allergic reaction or adverse reaction to cannabis is exclusionary.
* History of respiratory illness or current respiratory illness
* Currently enrolled in another research protocol
* Not using a contraceptive method (hormonal or barrier methods)
* Insensitivity to the cold water stimulus of the Cold Pressor Test
* Any disorders that might make cannabis administration hazardous are exclusionary, as determined by the evaluating physician

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Prospective research participants will be healthy, occasional (cannabis use biweekly to ≤ 3 day per week) cannabis-using men and non-pregnant and non-lactating women who will be evaluated for participation according to the following inclusion/exclusion criteria.
Enrollment: 20 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Analgesia | 7 hours
  Pain threshold and pain tolerance assessed with the Cold Pressor Test - time to report first feeling pain (0-180 seconds) and remove the hand from the cold water (0-180 seconds). Increased duration means increased pain tolerance and pain threshold.
Appetite stimulation | 7 hours
  Subjective ratings of hunger assessed with a visual analog scale (0-100 mm; 0 mm = no effect, 100 mm = maximum possible effect). Higher ratings indicate higher ratings of hunger / appetite stimulation.
Abuse liability | 7 hours
  Subject ratings of "Good Drug Effect" as measured using a visual analog scale (0-100 mm; 0 mm = no effect, 100 mm = maximum possible effect). Higher ratings indicate higher ratings of abuse liability.

SECONDARY OUTCOMES:
Subjective ratings of intoxication | 7 hours
  Subject ratings of "High" as measured using a visual analog scale (0-100 mm; 0 mm = no effect, 100 mm = maximum possible effect). Higher ratings indicate higher ratings of intoxication.
Subjective ratings of pain | 7 hours
  Subject ratings of Painfulness and Bothersomeness of the Cold Pressor Test. Scale is from 0 (Not painful / bothersome at all) to 10 (The most painful / bothersome feeling imaginable), higher ratings indicate greater painfulness and bothersomeness.

CONTACTS AND LOCATIONS:
Overall Officials: Ziva D Cooper, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No